CLINICAL TRIAL: NCT07244822
Title: A Randomized Controlled Trial Comparing the Effectiveness of Dexmedetomidine Versus Sufentanil on Cerebral Oxygen Saturation in Patients With Traumatic Brain Injury (DESTIN Trial)
Brief Title: Effectiveness of Dexmedetomidine Versus Sufentanil on Cerebral Oxygen Saturation in Patients With Traumatic Brain Injury
Acronym: DESTIN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitas Jenderal Soedirman (Other)
Collaborators: RS Prof. Dr. Margono Soekardjo Purwokerto (Unknown)
Responsible Party: Principal Investigator, MM Rudi Prihatno, Consultant Neuroanesthesiologist and Dean, Faculty of Medicine, Universitas Jenderal Soedirman, Universitas Jenderal Soedirman
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Jenderal Soedirman University; 079/KEPK/PE/VI/2025 (Registry Identifier: KEPK Faculty of Medicine Unsoed)
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Traumatic Brain Injury; Cerebral Oxygen Saturation; NIR Spectroscopy
Keywords: Traumatic Brain Injury; RSO2; NIRS; Dexmedetomidine; Sufentanil
MeSH Terms: conditions — Brain Injuries, Traumatic | interventions — Dexmedetomidine; Sufentanil

STUDY DESIGN:
Intervention Model Description: This is a randomized, controlled, parallel-group clinical trial designed to compare the effectiveness of dexmedetomidine versus sufentanil on cerebral oxygen saturation in patients with traumatic brain injury (TBI) undergoing surgery under general anesthesia. Participants will be randomly assigned in a 1:1 ratio into two intervention groups. The dexmedetomidine group will receive an induction dose of 1 µg/kg followed by maintenance at 0.3 µg/kg/hour, while the sufentanil group will receive an induction dose of 0.2 µg/kg followed by maintenance at 0.2 µg/kg/hour.
  Cerebral oxygen saturation will be continuously monitored using NIRS at baseline and postoperatively. The study aims to determine whether dexmedetomidine provides superior preservation of cerebral oxygenation compared to sufentanil. Randomization will be performed performed using simple random allocation (drawing method). Data will be analyzed based on intention-to-treat principles to compare changes in rSO₂ between two groups.
Who Masked: Participant, Care Provider
Masking Description: This study uses a double-blind design. Both the participants and the principal investigator are blinded to group allocation. Randomization is performed using a simple draw method assigning subjects to Group A or Group B. The anesthetic drugs (dexmedetomidine or sufentanil) are prepared and administered by an anesthesia team member who is not involved in data collection or outcome assessment. The study drugs are provided in identical, unlabeled syringes to ensure blinding. Neither the patients nor the investigator responsible for data recording and analysis will know which drug is administered until the study is completed and unblinding is authorized.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Active Comparator): Patients receive dexmedetomidine 1 µg/kg IV bolus for induction, followed by maintenance infusion at 0.3 µg/kg/h, combined with thiopental 5 mg/kg, rocuronium 0.6 mg/kg, and sevoflurane 1-1.5 vol% for maintenance anesthesia.
  Interventions: Drug: Dexmedetomidine
- Sufentanil group (Active Comparator): Patients receive sufentanil 0.2 µg/kg IV bolus for induction, followed by maintenance infusion at 0.2 µg/kg/h, combined with thiopental 5 mg/kg, rocuronium 0.6 mg/kg, and sevoflurane 1-1.5 vol% for maintenance anesthesia.
  Interventions: Drug: Sufentanil

INTERVENTIONS:
Drug: Dexmedetomidine — Dexmedetomidine administered as a 1 µg/kg IV bolus over 10 minutes before induction, followed by continuous infusion at 0.3 µg/kg/h during surgery. Used for anesthesia maintenance in patients with traumatic brain injury.
  Other Names: Neodex; Dexmeto
  Arms: Dexmedetomidine group
Drug: Sufentanil — Sufentanil administered as a 0.2 µg/kg IV bolus before induction, followed by continuous infusion at 0.2 µg/kg/h during surgery. Used for anesthesia maintenance in patients with traumatic brain injury.
  Other Names: Sufenta
  Arms: Sufentanil group

SUMMARY:
This randomized controlled clinical trial aims to evaluate the effectiveness of dexmedetomidine compared with sufentanil on cerebral oxygen saturation in patients with traumatic brain injury (TBI) undergoing surgery under general anesthesia. Cerebral oxygen saturation (rSO₂) will be monitored using Near-Infrared Spectroscopy (NIRS) to assess the impact of both anesthetic regimens on cerebral oxygenation and hemodynamic stability.

Patients meeting the inclusion criteria will be randomly assigned into two groups (1:1 ratio) using a simple random draw method.

Group A will receive dexmedetomidine 1 µg/kg for induction, thiopental 5 mg/kg, and rocuronium 0.6 mg/kg, followed by maintenance with dexmedetomidine 0.3 µg/kg/hour and sevoflurane 1-1.5 vol%.

Group B will receive sufentanil 0.2 µg/kg for induction, thiopental 5 mg/kg, and rocuronium 0.6 mg/kg, followed by maintenance with sufentanil 0.2 µg/kg/hour and sevoflurane 1-1.5 vol%. Both groups will receive intravenous paracetamol 1 g for analgesia at the end of surgery.

All patients will remain intubated postoperatively and will be transferred to the Intensive Care Unit (ICU) for monitoring. NIRS probes will be placed bilaterally on the cleaned frontal regions to measure rSO₂ values preoperatively, intraoperatively, and postoperatively at 60 and 120 minutes after intervention.

Postoperative analgesia will consist of dexmedetomidine 0.3 µg/kg/hour with paracetamol 1 g every 8 hours in the dexmedetomidine group, and sufentanil 0.1 µg/kg/hour with paracetamol 1 g every 8 hours in the sufentanil group.

Clinical and hemodynamic parameters will be recorded throughout the perioperative period.

Data will be analyzed to compare cerebral oxygen saturation changes between the two groups, aiming to determine whether dexmedetomidine provides superior cerebral oxygenation compared with sufentanil in patients with traumatic brain injury undergoing neurosurgical procedures.

DETAILED DESCRIPTION:
Traumatic brain injury (TBI) is a major cause of morbidity and mortality worldwide, often leading to secondary brain injury caused by hypoxia, ischemia, and impaired cerebral autoregulation. During anesthesia and surgery, maintaining adequate cerebral oxygenation is critical to prevent secondary neuronal damage. Cerebral oxygen saturation, measured by Near-Infrared Spectroscopy (NIRS), provides a continuous and noninvasive assessment of regional cerebral oxygenation (rSO₂), reflecting the balance between oxygen delivery and consumption in brain tissue.

Opioids such as sufentanil have traditionally been used to provide analgesia and hemodynamic stability during anesthesia in neurosurgical patients. However, opioid-related adverse effects, including respiratory depression, hypercapnia, and potential increases in intracranial pressure, raise concerns in patients with brain injury. Dexmedetomidine, a selective α₂-adrenergic receptor agonist, has sedative, analgesic, and sympatholytic properties without significant respiratory depression. It is known to reduce cerebral metabolic rate and intracranial pressure while maintaining cerebral perfusion, making it a potentially advantageous agent in neuroanesthesia.

This randomized controlled clinical trial aims to compare the effectiveness of dexmedetomidine versus sufentanil on cerebral oxygen saturation in patients with traumatic brain injury undergoing surgery. The hypothesis is that dexmedetomidine provides better maintenance of cerebral oxygenation, as measured by NIRS, compared to sufentanil under equivalent anesthetic conditions.

Eligible participants will be randomly allocated into two groups (1:1 ratio). The dexmedetomidine group will receive an induction dose of dexmedetomidine 1 µg/kg, thiopental 5 mg/kg, and rocuronium 0.6 mg/kg, followed by maintenance with dexmedetomidine 0.3 µg/kg/hour and sevoflurane 1-1.5 vol%. The sufentanil group will receive sufentanil 0.2 µg/kg, thiopental 5 mg/kg, and rocuronium 0.6 mg/kg, followed by sufentanil 0.2 µg/kg/hour and sevoflurane 1-1.5 vol%. All patients will receive intravenous paracetamol 1 g at the end of surgery for postoperative analgesia.

Postoperatively, patients will remain intubated and monitored in the Intensive Care Unit (ICU). Cerebral oxygen saturation (rSO₂) will be recorded using NIRS probes placed bilaterally on the frontal region before induction, during surgery, and at 60 and 120 minutes post-intervention in the ICU. Additional hemodynamic parameters including heart rate, mean arterial pressure, and oxygen saturation will also be recorded.

The primary outcome of this study is the change in cerebral oxygen saturation (rSO₂) between the two groups. Data obtained will be analyzed statistically to determine the comparative effectiveness of dexmedetomidine and sufentanil in maintaining optimal cerebral oxygenation during neurosurgical anesthesia in patients with traumatic brain injury. Findings from this study are expected to provide evidence-based recommendations for optimizing anesthetic management in neurotrauma cases, minimizing secondary brain injury, and improving patient outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-65 years diagnosed with traumatic brain injury (TBI) requiring surgical intervention under general anesthesia.
* Classified as ASA Physical Status I-III.
* Undergoing elective or emergency craniotomy at RSUD Prof. Dr. Margono Soekarjo Purwokerto.
* Provide informed consent (patient or legal representative).

Exclusion Criteria:

* Patients with severe cardiovascular instability (e.g., shock, uncontrolled arrhythmia).
* History of allergy or hypersensitivity to dexmedetomidine or sufentanil.
* Severe hepatic or renal impairment.
* Pregnant or lactating women.
* Glasgow Coma Scale ≤ 8 before induction.
* Refusal of participation or incomplete consent.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-31 (Actual); Study Completion 2025-08-31 (Actual)

PRIMARY OUTCOMES:
Cerebral oxygen saturation (rSO₂) measured by Near-Infrared Spectroscopy (NIRS) | Baseline (before induction), 60 minutes after surgery, and 120 minutes after surgery.
  Measurement of regional cerebral oxygen saturation (rSO₂) using Near-Infrared Spectroscopy (NIRS) placed bilaterally on the forehead. The mean rSO₂ values during and after anesthesia will be compared between the dexmedetomidine and sufentanil groups to assess cerebral oxygenation before and after surgery in traumatic brain injury patients.

CONTACTS AND LOCATIONS:
Overall Officials: Rudi Prihatno, Sp.An-Ti-KNA, Principal Investigator — Universitas Jenderal Soedirman
Locations (1):
- RSUD Prof. Margono Soekarjo, Purwokerto, Central Java, Indonesia

IPD SHARING:
Plan to Share IPD: No
The individual participant data (IPD) will not be shared because of institutional privacy policy and ethical considerations involving patient data from RSUD Prof. Dr. Margono Soekarjo Purwokerto.